CLINICAL TRIAL: NCT03174275
Title: Multimodality Therapy With Induction Carboplatin/Nab-Paclitaxel/Durvalumab Followed by Surgical Resection and Risk-adapted Adjuvant Therapy for the Treatment of Locally-Advanced and Surgically Resectable Squamous Cell Carcinoma of the Head and Neck
Brief Title: Carboplatin, Nab-Paclitaxel, Durvalumab Before Surgery and Adjuvant Therapy in Head and Neck Squamous Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: AstraZeneca (Industry); Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1621
Record Dates: First submitted 2017-05-26; First posted 2017-06-02 (Actual); Results first posted 2023-02-08 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Carcinoma, Squamous Cell; Oral Cancer; Oropharynx Cancer; Larynx Cancer; Lip Cancer; Esophageal Cancer
Keywords: squamous cell carcinoma of the head and neck (SCCHN); durvalumab; neoadjuvant induction; post-operative treatment
MeSH Terms: conditions — Carcinoma, Squamous Cell; Mouth Neoplasms; Oropharyngeal Neoplasms; Laryngeal Neoplasms; Lip Neoplasms; Esophageal Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — durvalumab; Carboplatin; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Cisplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low Risk (Experimental): Part 1- Patients receive 6 weeks of induction chemotherapy comprised of weekly cycles of carboplatin dosed to an Area Under the Curve (AUC2) and nab-paclitaxel 100 mg/m2 X 6 cycles in combination with durvalumab 750 mg administered once every two weeks for 5 cycles (D1 of weeks 1, 3, 5, 7, and 9).
  Part 2- Within a 2-6 week window post induction, tumor imaging will be followed by surgical resection.
  Part 3- patients receive adjuvant durvalumab (750 mg) once every two weeks x 3 cycles
  Interventions: Drug: Durvalumab; Drug: Carboplatin; Drug: Nab-paclitaxel; Procedure: Surgical resection
- Medium Risk (Experimental): Part 1- Patients receive 6 weeks of induction chemotherapy comprised of weekly cycles of carboplatin dosed to an Area Under the Curve (AUC2) and nab-paclitaxel 100 mg/m2 X 6 cycles in combination with durvalumab 750 mg administered once every two weeks for 5 cycles (D1 of weeks 1, 3, 5, 7, and 9).
  Part 2- Within a 2-6 week window post induction, tumor imaging will be followed by surgical resection.
  Part 3- patients receive ipsilateral involved field radiation concurrent with weekly cisplatin 30mg/m2. Once chemoradiotherapy is complete these patients will receive durvalumab 750 mg every two weeks for 3 cycles.
  Interventions: Drug: Durvalumab; Drug: Carboplatin; Drug: Nab-paclitaxel; Drug: Cisplatin; Procedure: Surgical resection; Radiation: IMRT
- High Risk (Experimental): Part 1- Patients receive 6 weeks of induction chemotherapy comprised of weekly cycles of carboplatin dosed to an Area Under the Curve (AUC2) and nab-paclitaxel 100 mg/m2 X 6 cycles in combination with durvalumab 750 mg administered once every two weeks for 5 cycles (D1 of weeks 1, 3, 5, 7, and 9).
  Part 2- Within a 2-6 week window post induction, tumor imaging will be followed by surgical resection.
  Part 3- All patients will be treated with intensity modulation radiation therapy (IMRT) concurrent with weekly cisplatin 30mg/m2 or other standard of care chemoradiotherapy regimen.Once chemoradiotherapy is complete these patients will receive durvalumab 750 mg every two weeks for 3 cycles.
  Interventions: Drug: Durvalumab; Drug: Carboplatin; Drug: Nab-paclitaxel; Drug: Cisplatin; Procedure: Surgical resection; Radiation: IMRT

INTERVENTIONS:
Drug: Durvalumab — Subjects will receive durvalumab, 750 mg every 2 weeks by IV infusion over approximately 1 hour (± 5 minutes).
  Other Names: MEDI4736
Drug: Carboplatin — Carboplatin is commercially available and approved by the US FDA for use in patients with ovarian cancer.
  Other Names: Paraplatin
Drug: Nab-paclitaxel — Nab-paclitaxel is commercially available and approved by the US Food and Drug Administration (FDA) for use in patients with metastatic breast cancer, metastatic pancreatic cancer, and for the treatment of locally advanced or metastatic NSCLC.
  Other Names: Abraxane
Drug: Cisplatin — Cisplatin is commercially available and approved by the US Food and Drug Administration (FDA) for the treatment of advanced bladder, ovarian and testicular cancer. It has been widely studied in a variety of solid tumor types.
  Arms: High Risk; Medium Risk
Procedure: Surgical resection — Surgical therapy will be at the discretion of the treating surgeon per standard of care.
Radiation: IMRT — "involved field radiation" will refer to areas demonstrated to harbor disease on pathology, and not elective areas
  Other Names: Intensity-modulated radiation therapy
  Arms: High Risk; Medium Risk

SUMMARY:
Participants in this study have a type of cancer called squamous cell carcinoma of the head and neck (SCCHN). Their SCCHN has spread around the area where the cancer first started. This is called locally-advanced SCCHN. These participants are eligible for surgery.

Previous research with a similar therapy regimen resulted in high rates of cancer shrinkage, high rates of avoiding radiation and its side effects, high cure rate and good quality of life. Radiation can be very toxic. The purpose on this study is to try to avoid radiation. If the participants are not on this study they would be receiving radiation as it is standard treatment of their cancer. In the last study with a similar regimen, about a third of cancers had a pathologic complete response with the first part of the study. This means that the chemotherapy had killed the cancer. The investigators are trying to improve the regimen further with a goal of increasing this rate of complete response to the first part of therapy. The investigators also hope that by improving results in the first part, that more people will be cured and that long term quality of life (especially speech and swallowing) will be improved, both compared to standard therapies and to the last study. Doctors do not know how this therapy will effect the participants. There is no guarantee that this study will benefit the participants.

The prior study used a combination of chemotherapy consisting of carboplatin, paclitaxel and a third targeted anti-cancer drug. In this study the investigators are testing the combination of carboplatin, nano-albumin bound paclitaxel and durvalumab. Nano-albumin bound paclitaxel has been shown to be more active against other types of squamous cancers than regular paclitaxel. It is FDA approved for squamous lung cancer, but experimental for head and neck cancer. Durvalumab is an experimental drug that uses the body's own immune system to fight the cancer. Doctors hope that combining Durvalumab with 2 chemotherapy drugs will be effective in treating SCCHN. Durvalumab on its own has been studied in patients with SCCHN and initial results have shown that some subjects' cancer has responded to it.

The purpose of this study is to test a combination of chemotherapy to hopefully both increase the number of subjects that respond to therapy while also decreasing the number of side effects that subjects experience.

DETAILED DESCRIPTION:
STUDY OBJECTIVES

Primary Objective:

Estimate the pathologic complete response rate (pCRR) after induction chemotherapy with carboplatin, nab-paclitaxel, and durvalumab in previously untreated stage III and IV SCCHN amenable to surgical resection

Secondary Objectives:

* Report the clinical complete response rate (cCRR) and clinical response rate (cRR) following induction chemotherapy
* Estimate the percent of patients who have a change in estimated risk level. Prior to induction, this will be assessed clinically (by imagining and physical exam). Post induction, this will be assessed by surgical pathology report
* Estimate the overall survival (OS) and progression free survival (PFS) associated with 3 part therapy consisting of induction chemotherapy, surgery and risk-adapted use of chemoradiation
* Characterize the toxicity profile associated with both induction therapy and total 3 part therapy consisting of induction chemotherapy, surgery and risk-adapted use of chemoradiation

Translational/Exploratory Objectives:

* Correlative studies will evaluate cellular correlates of response and changes in the tumor microenvironment across therapy
* Explore correlation between measures of clinical response to induction chemotherapy and long term outcomes (PFS and OS) and compare them to pathologic measures of response (pCRR)

PROCEDURES This is a single-arm, nonrandomized phase II trial consisting of 3 parts. After informed consent and screening, pre-induction, risk levels will be assessed clinically, by a combination of physical exam and imaging.

Part 1: All patients will then receive 6 weeks of induction chemotherapy in Part 1 comprised of weekly cycles of carboplatin and nab-paclitaxel for 6 cycles in combination with durvalumab administered once every two weeks for 5 cycles (Day 1 of the weeks 1, 3, 5, 7, and 9).

Part 2: Within a 1-4 the week window post induction, tumor imaging will be followed by surgical resection.

Part 3: After surgery, patients will be stratified into one of 3 risk categories based on their disease pathology, assigned a treatment group based on their risk. Low risk patients with receive durvalumab once every two weeks for 3 cycles, while medium risk or high risks groups will receive concurrent chemoradiation therapy followed by durvalumab once every two weeks for 3 cycles.

Follow up After completion of study therapy (which will vary by study arm) patients will be evaluated every three months during follow up for progression over a period of 18 months. Each follow up visit will include physical examination, CT or MRI imaging of the neck. Chest imaging will be obtained (or not) as indicated by standard of care. After the first 18 months, patients will be followed-up per standard of care, with documentation in the case report form (CRF) limited to progression and survival noted at their standard of care visits. If a patient should move away or otherwise be lost to in-person follow up but is amenable to telephone follow up, this will be permitted during the standard of care follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated, histologically proven, surgically resectable primary squamous cell carinoma of the head and neck, stage III or IV (HPV positive or negative non-metastatic disease). SCCHN of unknown primary is excluded. SCCHN of the oral cavity is allowed*. Unambiguously squamous Epstein-Barr virus (EBV)-negative nasopharynx cancer will be excluded nor will unambiguously squamous cancers of the skull base that are clearly surgically resectable and clearly squamous. Squamous skin cancer occurring in the head/neck region will not be eligible nor will EBV+positive nasopharynx cancer. (*Note: Induction chemotherapy is not considered standard therapy for SCCHN of the oral cavity and participation on this trial will lead to a delay in time to definitive, potentially curative therapy i.e., surgery).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Measurable disease as per RECIST 1.1
* Age greater than or equal to 18 at time of study entry
* Adequate bone marrow function as demonstrated by:

  * Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3
  * Hgb > 10 g/dL (use of transfusion to reach this threshold prior to study initiation is acceptable)
  * Platelet count ≥ 100,000/mm3
* Adequate hepatic and renal function as demonstrated by:

  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x upper limit of normal (ULN);
  * Total serum bilirubin ≤1.5 x ULN
  * Creatinine clearance (CrCL) > 40 mL/min as measured via Cockcroft-Gault

    * Males: Creatinine CL (mL/min) = (Weight (kg) x (140 - Age))/(72 x serum creatinine (mg/dL))
    * Females: Creatinine CL (mL/min) = (Weight (kg) x (140 - Age))/(72 x serum creatinine (mg/dL)) x 0.85
* Negative serum β human chorionic gonadotropin (β-hCG) pregnancy test within 72 hours of day 1 of induction chemotherapy in women of child-bearing potential.
* All males and females of childbearing potential must agree to use adequate contraception during the study. Adequate contraception is defined as any medically recommended method (or combination of methods) as per standard of care. Females of non-childbearing potential are those who are postmenopausal greater than 1 year or who have had a bilateral tubal ligation or hysterectomy or bilateral oophorectomy. See section 4.13 for list of acceptable methods of contraception.
* Signed an institutional review board (IRB)-approved informed consent and HIPAA authorization.
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Subjects must agree to allow use of any pre-treatment tissue remaining after definitive diagnosis is made (ie, archival and or fresh tissue) for research purposes. In addition, subjects must consent to allow use of their residual post-operative tissue for research purposes.

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to staff at the study site) or previous enrollment in the present study.
* Any metastatic disease.
* Known history of previous clinical diagnosis of tuberculosis.
* History and/or confirmed pneumonitis.
* Low-risk HPV+ disease of the oropharynx, defined as meeting all of the following criteria:

  * Patients with known HPV+ by fluorescence in situ hybridization (FISH) and/or p16
  * Smoking history ≤ 10 pack years
  * Stage T1-2N0-2b, T3N0
* Not considered eligible for any of the chemotherapy agents included in the induction regimen.
* Current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, or stable chronic liver disease per investigator assessment).
* Major surgery within 28 days prior to day 1 of study treatment from which the patient has not completely recovered.
* Receiving any investigational agent currently or within 28 days or 5 half-lives of Day 1 of treatment on this study, whichever is shorter.
* Active, serious infection, medical, or psychiatric condition that would represent an inappropriate risk to the patient or would likely compromise achievement of the primary study objective, including unstable angina, serious uncontrolled cardiac arrhythmia, uncontrolled infection, or myocardial infarction ≤ 6 months prior to study entry.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis, Crohn's disease], diverticulitis with the exception of a prior episode that has resolved or diverticulosis, celiac disease, irritable bowel disease, or other serious gastrointestinal chronic conditions associated with diarrhea; systemic lupus erythematosus; Wegener's syndrome [granulomatosis with polyangiitis]; myasthenia gravis;; rheumatoid arthritis; hypophysitis, uveitis; etc) within the past 2 years prior to the start of treatment. [Note: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded]
* Known mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Frediricia's Correction. (Note that ECG is not required for study entry and is not part of study procedures).
* Other prior or concomitant malignancies with the exception of:

  * Non-melanoma skin cancer
  * In-situ malignancy
  * Low-risk prostate cancer after curative therapy
  * Other cancer for which the patient has been disease free for ≥ 5 years before the first dose of study drug and of low potential risk for recurrence.
* Any concurrent chemotherapy, investigational product, biologic or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g. hormone replacement therapy) is acceptable.
* Current or prior use of immunosuppressive medication within 14 days prior to the first dose of durvalumab. The following are exceptions to this criterion: intranasal, inhaled, topical or local steroid injections (eg. intra-articular injection); steroids as premedication for hypersensitivity reactions; systemic corticosteroid at physiologic doses not to exceed 10mg/day of prednisone or equivalent.[Note: If systemic corticosteroids are part of the treatment regimen for the indication under study, the systemic corticosteroid is permitted].
* Known human immunodeficiency virus (HIV), hepatitis C virus (HCV) or evidence of active hepatitis B virus (HBV).
* History of hypersensitivity to durvalumab or any excipient.
* Receipt of live attenuated vaccination within 30 days prior the first dose of durvalumab [Note: If a vaccine is part of the treatment regimen for the indication under study, the vaccine is permitted].
* Female subjects who are pregnant, breast-feeding or female patients of reproductive potential who are not employing an effective method of birth control from starting dose of study medications (Cycle 1 Day 1), including dosing interruptions through 90 days after receipt of the last dose of durvalumab. Refrain from egg cell donation while taking durvalumab and for at least 90 days after the last dose of durvalumab.
* Male subjects who are not employing an effective method of birth control from starting dose of study medications (Cycle 1 Day 1), including dosing interruptions through 6 months after receipt of study treatment. Male subjects should agree to refrain from sperm donation while taking study treatment and for at least 6 months after the last dose of nab-paclitaxel and at least 90 days after the last dose of durvalumab. Should a female partner of a male patient become pregnant or suspect she is pregnant while participating in the study, he should inform his treating physician and the female partner should call her physician immediately.
* Any previous treatment with a programmed cell death protein 1 (PD-1) or programmed death-ligand 1 (PD-L1) inhibitor, including durvalumab.
* History of primary immunodeficiency.
* History of organ transplant.
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results (eg, uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent).
* Patients with known contraindications to radiotherapy including inherited syndromes associated with hypersensitivity to ionizing radiation (e.g., Ataxia Telangiectasia, Nijmegen Breakage Syndrome).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2027-02-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jared Weiss, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - Lineberger Comprehensive Cancer Center at University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trial — https://unclineberger.org/patientcare/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 12/19/2017 through 11/09/2021 at 4 cancer centers in the United States.
Pre-assignment Details: A total of 44 participants consented, but 5 were deemed to be ineligible, and 39 subjects enrolled in the study; 37 out of 39 subjects completed neoadjuvant therapy, and 2 subjects were off the treatment due to toxicity; 35 out of 37 subjects underwent surgery at study centers, one subject had surgery elsewhere, and one subject declined the surgery. Subjects received adjuvant therapy based on surgical pathology results and treatment progress was submitted separately.
Groups:
- All Study Subjects: Subjects received at least one dose of study treatment
Period: Overall Study (Until End of Surgery)
Arm/Group | All Study Subjects
Started | 39
Completed | 25
Not Completed | 14
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 9
Not completed — Lack of Efficacy | 1
Period: Adjuvant Chemotherapy
Arm/Group | All Study Subjects
Started | 21 (The participants were prescribed adjuvant chemotherapy based on the surgical pathology report included.)
Completed | 13
Not Completed | 8
Not completed — Withdrawal by Subject | 6
Not completed — Progression | 1
Not completed — Adverse Event | 1
Period: Adjuvant Durvalumab
Arm/Group | All Study Subjects
Started | 35 (The participants were prescribed adjuvant durvalumab based on the surgical pathology report included.)
Completed | 25
Not Completed | 10
Not completed — Withdrawal by Subject | 6
Not completed — Progression | 1
Not completed — Adverse Event | 3
Period: Adjuvant Radiotherapy
Arm/Group | All Study Subjects
Started | 21 (The participants were prescribed adjuvant radiotherapy based on the surgical pathology report included.)
Completed | 14
Not Completed | 7
Not completed — Withdrawal by Subject | 5
Not completed — Progression | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: This study protocol requires the same neoadjuvant therapy and surgery for all subjects. Adjuvant treatment is assigned based on the risk group. The primary outcome measure is the complete pathologic response that is defined by the surgical pathology report. Complete pathologic response is not related to adjuvant therapy.
Groups:
- All Subjects: All subjects received at least one dose of study treatment, from any of the arms (low risk, medium risk, and high risk). This study protocol requires the same neoadjuvant therapy and surgery for all subjects. Adjuvant treatment is assigned based on the risk group. Adjuvant treatment arms were not randomized. Therefore, baseline characteristics were reported based on the whole group.
Arm/Group | All Subjects
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 32
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response Rate (pCRR) After Induction Chemotherapy With Carboplatin, Nab-paclitaxel, and Durvalumab in Previously Untreated Stage III and IV SCCHN Amenable to Surgical Resection
Description: The pCRR was assessed via surgical pathology report. Pathologic complete response will require no viable cancer cells on the surgical pathology report after neoadjuvant treatment with carboplatin, nab-paclitaxel, and durvalumab. This study protocol requires the same neoadjuvant therapy and surgery for all subjects. The primary outcome measure is the complete pathologic response defined by the surgical pathology report and is unrelated to adjuvant therapy.
Time Frame: After surgery (approximately 8-12 weeks after start of study treatment)
Population: Subjects received treatment in 4 cancer centers in the United States.
Measure: Count of Participants; unit: Participants
Groups:
- Pathologic Complete Response: All subjects received neoadjuvant chemotherapy and underwent surgery, and histopathological analyses were completed.
Arm/Group | Pathologic Complete Response
Number analyzed (Participants) | 35
Participants
  Pathologic complete response was achieved | 10
  Pathologic complete response was not achieved | 25

2. Secondary Outcome: Clinical Complete Response Rate and (cCRR) and Clinical Response Rate (cRR) Following Induction Chemotherapy
Description: Clinical complete response rate and clinical response rate (CR + PR) associated with induction chemotherapy will be estimated using RECIST 1.1.
Time Frame: 1-4 weeks post induction chemotherapy
Reporting Status: Not Posted

3. Secondary Outcome: Percent of Patients Who Have a Change in Estimated Risk Level
Description: Risk level pre-induction will be based on physical examination and imaging and will be defined and documented in electronic Case Report Forms (eCRF) prior to the initiation of induction therapy. Post-induction risk level will be determined based on pathologic evaluation of surgical specimen.
Time Frame: After surgery (approximately 8-12 weeks after start of study treatment)
Reporting Status: Not Posted

4. Secondary Outcome: Progression Free Survival (PFS) Associated With 3 Part Therapy Consisting of Induction Chemotherapy, Surgery and Risk-adapted Use of Chemoradiation
Description: PFS will be defined as the time from day 1 of study treatment until progression per RECIST 1.1
Time Frame: 5 years
Reporting Status: Not Posted

5. Secondary Outcome: Overall Survival (OS) Associated With 3 Part Therapy Consisting of Induction Chemotherapy, Surgery and Risk-adapted Use of Chemoradiation
Description: Overall survival will be defined as the time from day 1 of study treatment until death from any cause
Time Frame: 5 years
Reporting Status: Not Posted

6. Secondary Outcome: Toxicity Profile Associated With Both Induction Therapy and Total 3 Part Therapy Consisting of Induction Chemotherapy, Surgery and Risk-adapted Use of Chemoradiation
Description: Safety associated with both induction alone and with 3 part therapy consisting of induction chemotherapy, surgery and risk-adapted use of chemoradiation will be assessed via the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE v4.03)
Time Frame: 90 days after the last dose of study treatment
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Cellular Correlates of Response and Changes in the Tumor Microenvironment Across Therapy
Description: Pre-treatment specimens will be studied for predictive markers of treatment response. Paired pre- and post-treatment specimens will be compared to assess for changes in the tumor micro-environment.
Time Frame: 8-12 weeks after the last dose of study treatment
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Correlation Between Measures of Clinical Response to Induction Chemotherapy and Long Term Outcomes (PFS and OS) and Compare Them to Pathologic Measures of Response (pCRR).
Description: as for outcome 7
Time Frame: 8-12 weeks after the last dose of study treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected from day one of the study drug administration to 30 days after completion of adjuvant treatment, up to 9 months.
Description: CTCAEv4
Groups:
- All Subjects: This study protocol requires the same neoadjuvant therapy and surgery for all subjects. Adjuvant treatment is assigned based on the risk group. Adjuvant treatment arms were not randomized. Therefore, Adverse Events were reported based on the whole group.
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/39
Serious Adverse Events (participants affected / at risk) | 9/39
Other Adverse Events (participants affected / at risk) | 38/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Subjects (N=39)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Endocrine disorders - Other, specify (Endocrine disorders) | 1
Dysphagia (Gastrointestinal disorders) | 3
General disorders and administration site conditions - Other, specify (General disorders) | 1
Lung infection (Infections and infestations) | 2
Sepsis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Tracheitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Glucose intolerance (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Subjects (N=39)
Anemia (Blood and lymphatic system disorders) | 37
Blood and lymphatic system disorders other (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 1
Heart failure (Cardiac disorders) | 1
Mitral valve disease (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Ear pain (Ear and labyrinth disorders) | 3
External ear pain (Ear and labyrinth disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 3
Tinnitus (Ear and labyrinth disorders) | 9
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 5
Blurred vision (Eye disorders) | 3
Eye disorders - Other, specify (Eye disorders) | 3
Flashing lights (Eye disorders) | 1
Floaters (Eye disorders) | 1
Photophobia (Eye disorders) | 1
Watering eyes (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Colitis (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 29
Diarrhea (Gastrointestinal disorders) | 19
Dry mouth (Gastrointestinal disorders) | 8
Dysphagia (Gastrointestinal disorders) | 7
Flatulence (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 8
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 14
Nausea (Gastrointestinal disorders) | 28
Oral hemorrhage (Gastrointestinal disorders) | 4
oral pain (Gastrointestinal disorders) | 15
Stomach pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 9
Chills (General disorders) | 3
Edema face (General disorders) | 1
Edema limbs (General disorders) | 4
Facial pain (General disorders) | 2
Fatigue (General disorders) | 36
Fever (General disorders) | 5
Flu like symptoms (General disorders) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 5
Localized edema (General disorders) | 1
Malaise (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 10
Autoimmune disorder (Hepatobiliary disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 3
Lung infection (Infections and infestations) | 1
Mucosal infection (Infections and infestations) | 5
Paronychia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 2
Skin infection (Infections and infestations) | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 11
Fracture (Injury, poisoning and procedural complications) | 1
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1
Wound complication (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 11
Alkaline phosphatase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 10
Blood bilirubin increased (Investigations) | 1
Cholesterol high (Investigations) | 1
Creatinine increased (Investigations) | 5
Lipase increased (Investigations) | 4
Lymphocyte count decreased (Investigations) | 27
Neutrophil count decreased (Investigations) | 27
Platelet count decreased (Investigations) | 23
Weight loss (Investigations) | 13
White blood cell decreased (Investigations) | 30
Anorexia (Metabolism and nutrition disorders) | 8
Dehydration (Metabolism and nutrition disorders) | 8
Hypercalcemia (Metabolism and nutrition disorders) | 5
Hyperglycemia (Metabolism and nutrition disorders) | 6
Hyperkalemia (Metabolism and nutrition disorders) | 9
Hypermagnesemia (Metabolism and nutrition disorders) | 4
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 11
Hypocalcemia (Metabolism and nutrition disorders) | 5
Hypokalemia (Metabolism and nutrition disorders) | 13
Hypomagnesemia (Metabolism and nutrition disorders) | 16
Hyponatremia (Metabolism and nutrition disorders) | 20
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Dizziness (Nervous system disorders) | 2
Dysarthria (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 15
Headache (Nervous system disorders) | 6
Memory impairment (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 7
Peripheral sensory neuropathy (Nervous system disorders) | 10
Seizure (Nervous system disorders) | 1
Stroke (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 11
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 14
Acute kidney injury (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 4
Sore throat (Respiratory, thoracic and mediastinal disorders) | 6
Alopecia (Skin and subcutaneous tissue disorders) | 27
Dry skin (Skin and subcutaneous tissue disorders) | 4
Nail discoloration (Skin and subcutaneous tissue disorders) | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 16
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 5
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 5
Hypotension (Vascular disorders) | 2
Superficial thrombophlebitis (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results should be deferred until published.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT03174275/Prot_SAP_000.pdf